CLINICAL TRIAL: NCT07264153
Title: Efficacy of High-Intensity Laser Therapy (HILT) in the Management of Isotretinoin-Induced Sacroiliitis: A Randomized Controlled Trial
Brief Title: Laser Therapy in the Isotretinoin-Induced Sacroiliitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uşak University (Other)
Responsible Party: Principal Investigator, Ali Yavuz Karahan, Professor, Uşak University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ayk 2025
Record Dates: First submitted 2025-11-23; First posted 2025-12-04 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Sacroilitis
Keywords: Laser Therapy; Isotretinoin; Sacroiliitis; Pain
MeSH Terms: conditions — Sacroiliitis; Pain | interventions — Laser Therapy; Exercise

STUDY DESIGN:
Intervention Model Description: A single-center, prospective, randomized, controlled, parallel-group trial with a 1:1 allocation ratio.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be blinded to the treatment allocation (assessor-blinded). The physiotherapist administering the therapy and participants and cannot be blinded due to the nature of the interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser Therapy Group (LTG) (Experimental): The treatment protocol comprised two distinct modes: the first being the administration of analgesic medication, and the second being biostimulation. For the analgesic mode, the laser was administered at an operating power of 10W, with the energy density set at 12J/cm2 across a surface area of 15cm2. The laser will applied in along the right and left sacroiliac joints for four minutes. The total energy delivered will 600 J. In the biostimulation mode, a laser with an operating power of 5 W will applied, generating an energy density of 120 J/cm2 across a surface area of 15 cm2 at the sacroiliac joint line for a duration of 10 minutes, resulting in a total energy output of 3,000 J.
  Application Technique: The applicator will be moved in a slow, circular, or grid pattern over the target area for 12 minutes.
  Interventions: Device: Laser Therapy; Other: Exercises for both groups
- Sham Therapy Group (STG) (Sham Comparator): Protocol and dosage: In all aspects, including the device's appearance, audible cues (e.g. timer beeps), treatment duration and the physical application of the probe to the skin, the sham protocol will be identical to the active protocol.
  Interventions: Other: Exercises for both groups

INTERVENTIONS:
Device: Laser Therapy — Protocol and dosage: Treatment will be applied directly over the painful sacroiliac joint(s). The treatment protocol comprised two distinct modes: the first being the administration of analgesic medication, and the second being biostimulation. For the analgesic mode, the laser was administered at an operating power of 10W, with the energy density set at 12J/cm2 across a surface area of 15cm2. The laser will applied in along the right and left sacroiliac joints for four minutes. The total energy delivered will 600 J. In the biostimulation mode, a laser with an operating power of 5 W will applied, generating an energy density of 120 J/cm2 across a surface area of 15 cm2 at the sacroiliac joint line for a duration of 10 minutes, resulting in a total energy output of 3,000 J.
  Application Technique: The applicator will be moved in a slow, circular, or grid pattern over the target area for 12 minutes.
  Arms: Laser Therapy Group (LTG)
Other: Exercises for both groups — Participants will be taught the supervised exercise programme. Sessions will be held three times per week on non-consecutive days. Each session will last approximately 45 minutes.
  The exercise programme was designed to address pain and dysfunction related to hypomobility and instability of the sacroiliac joint (SIJ). The intervention comprises a structured, progressive exercise regimen consisting of three sequential phases: 1) Gentle Movement and Relaxation, 2) Specific Self-Mobilisation and 3) Core and Stabilisation. The protocol will be delivered to participants in a standardised format, with progression based on individual tolerance and clinical milestones.

SUMMARY:
The clinical significance of this adverse effect lies in its impact on quality of life and the potential for misdiagnosis. The symptomatology can be severe enough to limit daily activities and may be mistakenly attributed to a primary rheumatic disease, leading to unnecessary long-term immunosuppressive therapy if the temporal link to isotretinoin is not identified. Therefore, a high index of suspicion is crucial for dermatologists, rheumatologists, and primary care physicians alike.

Aim: To compare the effectiveness of High-Intensity Laser Therapy (HILT) in reducing pain intensity, in patients diagnosed with Isotretinoin-Induced Sacroiliitis.

DETAILED DESCRIPTION:
Isotretinoin (13-cis-retinoic acid) is a highly effective retinoid derivative of vitamin A, renowned for its use in the treatment of severe, recalcitrant nodular acne. By significantly reducing sebum production, modulating follicular keratinization, and exerting anti-inflammatory effects, it has proven to be a transformative therapy for patients with conditions unresponsive to conventional treatments. However, its potent biological activity is accompanied by a well-documented and diverse profile of adverse effects, ranging from common mucocutaneous symptoms like xerosis and cheilitis to more serious concerns such as teratogenicity, psychiatric effects, and musculoskeletal complaints.

Among these musculoskeletal adverse events, sacroiliitis-the inflammation of one or both sacroiliac (SI) joints-has emerged as a significant, though potentially underrecognized, clinical entity. The sacroiliac joints, which connect the sacrum to the iliac bones of the pelvis, are a primary site for inflammatory processes seen in spondyloarthropathies (SpA) such as ankylosing spondylitis. The presentation of Isotretinoin-induced sacroiliitis often mirrors that of these idiopathic conditions, characterized by insidious-onset lower back pain, buttock pain, and stiffness that may improve with activity and worsen with rest. Morning stiffness is a common feature, and pain can often be referred to the groin or posterior thigh.

The pathophysiological mechanism linking isotretinoin to sacroiliitis remains incompletely elucidated but is a subject of active investigation. Retinoids are known to modulate the immune system, influencing the differentiation and proliferation of various immune cells. It is hypothesized that isotretinoin may disrupt the delicate balance between pro-inflammatory and anti-inflammatory cytokines, potentially triggering an inflammatory cascade in genetically predisposed individuals. This theory is supported by the observation that symptoms often resolve upon discontinuation of the drug and may recur upon re-challenge, satisfying important criteria for a causal relationship.

The clinical significance of this adverse effect lies in its impact on quality of life and the potential for misdiagnosis. The symptomatology can be severe enough to limit daily activities and may be mistakenly attributed to a primary rheumatic disease, leading to unnecessary long-term immunosuppressive therapy if the temporal link to isotretinoin is not identified. Therefore, a high index of suspicion is crucial for dermatologists, rheumatologists, and primary care physicians alike.

Aim: To compare the effectiveness of High-Intensity Laser Therapy (HILT) in reducing pain intensity, in patients diagnosed with Isotretinoin-Induced Sacroiliitis.

Secondary Objectives:

* To assess and compare the improvement in functional status and quality of life between the two intervention groups using validated questionnaires.
* To evaluate and compare the reduction in disease activity and inflammatory symptoms (e.g., morning stiffness, night pain) between the groups.
* To measure and compare the improvement in spinal mobility and specific sacroiliac joint provocation tests.
* To monitor the safety and adverse event profile of HILT in this patient population.

Study Design:

A single-center, prospective, randomized, controlled, parallel-group trial with a 1:1 allocation ratio. The outcome assessor will be blinded to the treatment allocation (assessor-blinded). The physiotherapist administering the therapy and participants and cannot be blinded due to the nature of the interventions.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 35 years.
* Receiving a stable dose of oral isotretinoin (e.g., 0.3-0.5 mg/kg/day) for at least one month.
* Diagnosis of sacroiliitis based on: Clinical symptoms: Persistent (≥4 weeks) lower back/buttock pain, morning stiffness >30 minutes, improvement with exercise. Positive physical findings: At least two positive sacroiliac joint provocation tests (e.g., FABER/Patrick's test, Gaenslen's test, Compression/Distraction test). Radiological confirmation (MRI): Active inflammation (bone marrow edema) on Short-Tau Inversion Recovery (STIR) sequences in one or both sacroiliac joints.
* A baseline pain intensity of ≥4 on the Visual Analog Scale (VAS 0-10 cm).

Exclusion Criteria:

* ankylosing spondylitis or other seronegative spondyloarthritis
* the presence of pregnancy
* the presence of any cancer
* the presence of multiple sclerosis

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2026-04-11 (Estimated); Study Completion 2026-05-11 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | will be performed at Baseline (T0), immediately after the 4-week intervention period (T1), and at a 1-month follow-up (T2) to assess sustainability.
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."
Pain Intensity | will be performed at Baseline (T0), immediately after the 4-week intervention period (T1), and at a 1-month follow-up (T2) to assess sustainability.
  Algometers are designed to quantify and document levels of tenderness via pressure pain threshold measurement and pain sensitivity via pressure pain tolerance measurement. The manual analogue algometer is a device that is utilised for the measurement of pressure that is applied manually. The device displays a real-time graph of the applied pressure on the analogue screen. The operator employs the use of guidance lines on the analogue screen, thereby enabling the precise application of pressure at the optimal rate. This facilitates the establishment of a highly standardised stimulus.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Y Karahan, Professor, Principal Investigator — Uşak University
Locations (1):
- University of Usak, Uşak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared. The investigators will publish the results in academic journals.